CLINICAL TRIAL: NCT02188407
Title: Phase 1 Study of Antiinflammatory Effect of Sevoflurane in Open Lung Surgery With One-Lung Ventilation
Brief Title: Inflammation After One Lung Ventilation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Iztok Potocnik, MD, MSC, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UKC-TOR-1
Record Dates: First submitted 2014-07-03; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Inflammation
Keywords: thoracotomy; one-lung ventilation (OLV); total intravenous anaesthesia (TIVA); volatile induced and maintained anaesthesia (VIMA); cytokines; interleukine (IL)
MeSH Terms: conditions — Inflammation | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane (Experimental): Sevoflurane group (S group)- The group anaesthesied with sevoflurane
  Interventions: Drug: Sevoflurane
- Propofol (Active Comparator): Propofol 4-6 mg/kg/h iv
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — MAC 3-5 V% during surgery
  Other Names: Sevorane
  Arms: Sevoflurane
Drug: Propofol — Propofol group (P group)- The group anaesthesied with propofol
  Arms: Propofol

SUMMARY:
The aim of the study was to prospectively investigate the influence of one-lung ventilation (OLV) on the inflammatory response and to identify possible antiinflammatory effects of the volatile anaesthetic sevoflurane.

Forty patients undergoing thoracic surgery with OLV were enrolled in this prospective, randomised study. The patients were randomly allocated into two groups to receive either propofol (Group P) or sevoflurane (Group S) for induction and maintenance of anaesthesia.

Inflammatory mediators (Interleukin 6 (IL6), Interleukin8 (IL8), Interleukin 10 (IL10), (C- reactive protein)CRP) were measured intra- and postoperatively.

Six hours after surgery oxygenation index (PaO2/FiO2) was calculated and chest X ray was taken and assessed.

The clinical outcome determinated by postoperative adverse events was assessed as the secondary endpoint.

DETAILED DESCRIPTION:
Lung injury is the main complication of open lung surgery and is associated with a very high mortality rate.

In 1984, Zeldin reported on ten patients with a complication that he referred to as postpneumonectomy pulmonary oedema (PLE). The complication is sometimes not easy to differentiate from acute respiratory distress syndrome (ARDS), defined by Bernard et al, because the patients may not fulfill all the ARDS criteria. The incidence of this so-called acute lung injury (ALI) after lobectomy is 1-7%. The mortality rate in patients with ARDS and ALI is 72% and 33%, respectively.

In patients undergoing lung resection, mechanical ventilation and surgery may induce alveolar and systemic inflammatory responses. One-lung ventilation (OLV) has become as a standard procedure for many interventions in thoracic surgery with a need for deflation of the lung to facilitate the surgical procedure. It is also the main cause of acute inflammatory response and is associated with ALI and ARDS. The inflammatory reaction produces injury to the lung endothelium. The loss of endothelium integrity causes increased protein leak into the alveolar fluid. The inflammatory reaction leads to other histological changes. These reactions during OLV have been reported by many investigators.

A number of studies have shown that sevoflurane attenuates cardiac ischaemia-reperfusion injury. These results have been lately transferred to lung surgery. Some studies have demonstrated that volatile anaesthetics sevoflurane, isoflurane and desflurane have an impact on ischaemic-reperfusion lung injury. These studies have confirmed the local alveolar, but not the systemic antiinflammatory effects of sevoflurane.

Studies to date have not evaluated long-lasting effects of anaesthetics administered intraoperatively.

Demonstrating the influence of volatile anaesthetics on the inflammatory response and the treatment outcome in patients undergoing open lung surgery with OLV is still a great challenge for thoracic anaesthesiologists.

The effects of sevoflurane on release of inflammatory markers has been addressed before, but the added value of our study is that we tested the systemic imunomodulatory effect of sevoflurane in combination with postoperative clinical outcome and adverse effects.

In the current study the following null hypothesis was tested: the administration of sevoflurane or propofol does not affect the systemic proinflammatory response after open lung surgery with OLV.

ANAESTHESIA REGIMEN All patients were given oral diazepam 5-10 mg (Apaurin, Krka, d.d.) one hour before surgery. On arrival in the operating room, they were randomly assigned to either Group P or Group S. Randomisation was done according to computer-generated order.

Antibiotic prophylaxis with intravenous (iv) cefazolin (Cefamezin, Krka, d.d.) 2g/100 ml 0.9% NaCl was used in all patients.

Standardised clinical monitoring devices were attached to all patients prior to induction of anaesthesia. For extended haemodynamic monitoring LiDCO plus system was used.

A thoracic epidural catheter was inserted at the T6-7 level. Anaesthesia induction in Group P was performed with propofol (Propoven, Fresenius Kabi) and in Group S with sevoflurane (Sevorane, Abbott Laboratories). Before intubation all patients received remifentanil (Ultiva, GlaxoSmithKline) and vecuronium (Norcuron, Organon).

All patients were intubated with a left-sided double-lumen endobronchial tube (Malinckrodt, with hook, 37-41 Charriere) and ventilated by volume-controlled ventilation, provided by a closed-circuit anaesthesia ventilator (Primus, Draeger, Luebeck, Germany). The tidal volume was set to 6 ml/kg. The peak inspiratory pressure was limited to 25 cm H2O. The fraction of inspired oxygen was adjusted to maintain oxyhaemoglobin saturation at greater than 96% (fraction of inspired oxygen 0.3 to 0.4 before OLV; fraction of inspired oxygen 0.6 to 0.7 during OLV, and the respiratory rate to keep the PaCO2 between 3.8-4.5 kPa. The positive end expiratory pressure (PEEP) was set to 5 cm H2O. Gas concentration and airway pressures were measured at the proximal end of the tube using ventilator-integrated functions. During OLV the tidal volume was set to 4 ml/kg and peak inspiratory pressure limited to 25 cm H2O. Other ventilation settings were maintained and PEEP was reduced to 3 cm H2O.

Anaesthesia was maintained with propofol in Group P (4-6 mg/kg/h) and with sevoflurane (V% 2-2.5) in Group S. The rate of remifentanil iv infusion was 0.3-0.5 mcg/kg/min in both groups. The depth of anaesthesia was measured by a bispectral index (BIS) monitor; BIS values were maintained at 40-60.

For haemodynamic management the following algorithm was used: continuous infusion of 0.9% NaCl 6 mL /kg for the first hour, followed by 2.5 ml /kg/h, if DO2I<600 ml/min/m2 and SVR> 800 and SVV > 10% 6% hydroxyethyl starch (Voluven, Fresenius Kabi) until SVV decreased under 10% ; if there was no improvement after 250 ml 6% HES-a, dobutamine (Inotop Torrex Pharma) 1-10 mcg/kg/min iv is introduced; if SVR < 800 dyn•s/cm5 then ephedrine (0.5% Efedrin, UMC Ljubljana Pharmacy) 5-10 mg iv was given. If the mean arterial pressure increases by more than 30% and the heart rate by more than 30% from baseline, the infusion of remifentanil is increased by 0.1mcg/kg/min.

At the end of the procedure, the action of muscle relaxants was reversed with neostigmine (Neostigmin-Actavis, Actavis) 2.5 mg and atropine (Atropinum sulfuricum, Nycomed) 1 mg iv. All patients were extubated in the operating theatre and then transferred to the recovery room.

POSTOPERATIVE MANAGEMENT After surgery, the patients stayed in the recovery room for one hour and were then transferred to the intensive care unit of the Department of Thoracic Surgery.

Standard postoperative monitoring generally used in these procedures was implemented. Haemodynamic monitoring using the LiDCO plus system was continued after surgery.

Oxygen titrated to the lowest level needed to achieve the target arterial oxygen saturation of 96%, was administered via a Venturi mask.

For postoperative haemodynamic management the following algorithm was implemented: continuous infusion of 0.9% NaCl 1 ml/kg/h , if oxygen delivery index (DO2I) was less than 600 ml/min/m2 and systemic vascular resistance (SVR) was higher than 800 dyn•s/cm5 infusion of 6% hydroxyethyl starch (Voluven, Fresenius Kabi), if no improvement occurs after 250 ml 6% HES, dobutamine (Inotop, Torrex Pharma) 1-10 mcg/kg/min was initiated, if SVR < 800 than ephedrine (0.5% Efedrin, Pharmacy UMC Ljubjana ) 5-10 mg iv was given.

In the recovery room, all patients received 10 ml of 0.5% levo-bupivacaine (Chirocaine, Abbott Laboratories) and the level of the epidural sensory block was tested. Postoperative analgesia was provided by infusion of 0.25 % levobupivacaine via an epidural catheter using a patient- controlled analgesia (PCA) pump. The infusion rate was 5 ml/h and lockout time 30 min. Hourly pain assessments using a visual analogue scale (VAS) were performed. Patients with VAS scores greater than 3 received a rescue analgetic piritramide 3 mg (Dipidolor, Johnson&Johnson) intravenously.

MEASUREMENTS The data recorded included demographic characteristics, time of surgery, time of OLV and DO2.

Arterial blood samples for the determinations of cytokines (IL 6, IL 8, IL 10), C-reactive protein (CRP) were drawn at the following time points: 1. before induction, 2. five minutes after the placement of the retractor, 3. 10 minutes after the beginning of OLV, 4. at the end of surgery, and 5. 6 hours after surgery. CRP was measured also 24 hours after the operation. For the analysis of serum CRP, IL 6, IL 8 and IL 10, blood samples were collected without additive. After centrifugation, serum samples were stored at -20 °C until analysis. Samples were analysed in one batch. CRP, IL 6, IL 8 and IL 10 were measured by a chemiluminescent immunometric assay (Immulite analyser; Simens Healthcare, Erlangen, Germany); a high-sensitivity method with a detection limit of 0.3 mg/L was used for measuring CRP.

Procalcitonin (PCT) levels were measured 6 and 24 hours after the operation. Chest X-rays were taken 6 hours after the procedure to evaluate the infiltration of the nonoperated lung. The following scoring was used: 0=no infiltration; 1=partly infiltrated; and 2= fully infiltratied.

The oxygenation index (ratio of partial arterial oxygen pressure to inspiratory fraction of oxygen =PaO2/FiO2) was calculated 6 hours after the procedure.

SECONDARY ENDPOINTS The clinical postoperative outcome was assessed as secondary endpoint based on adverse events. The following parameters were determined: prolonged antibiotics, diagnosed pneumonia, reintubation, systemic inflammatory response syndrome, sepsis, acute respiratory distress syndrome, acute renal failure, postoperative nausea and vomiting and death.

STATISTICAL ANALYSIS Statistical analysis were performed using the R software v 3 (R Development Core Team). All p-values reported are two-sided and the significance level was set at 5% (p < 0.05). Continuous variables are presented as mean ±SD.

Repeated measures ANOVA was used to identify differences in plasma CRP, IL6, IL8 and IL10 concentrations between the two study groups.

Based on authors' previous pilot study in 6 patients, to detect the significant difference of the IL 6 concentration with a significance level of 0.05 and a power of 80%, 16 patients in each group sufficed for the primary test. To compensate for withdrawals, 20 patients per group were included in the study.

Where appropriate t-test, Mann-Whitney tests and Chi-square test were also used.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-70 years
* American Society of Anaesthesiologists (ASA) physical status I-III
* elective open lobectomy with OLV

Exclusion Criteria:

* history of drug hypersensitivity
* drug addiction
* treatment with psychotropic drugs
* severe psychiatric and central nerve system diseases
* persistent tobacco abuse, autoimmune system diseases
* diabetes mellitus
* cardiac failure (New York Heart Association class greater than 2)
* clinically relevant obstructive and restrictive lung diseases (vital capacity or forced expiratory volume in 1s lover than 50% of the predicted values)
* pulmonary hypertension (mean pulmonary arterial pressure grater than 25 mmHg)
* pre-existing coagulation disorders
* history of treatment with immunosuppressant drugs in the 4 weeks before surgery
* Patient with evidence of pulmonary or systemic infections (C-reactive protein serum concentration greater than 5 mg/L, leucocytosis greater than 10.0 bioparticles/L or body temperature greater than 37 stC)
* perioperative blood derivatives, steroids or non-steroidal anti-inflammatory drug (NSAID)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-07; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
IL 6 | intraoperatively and 6 hours after surgery
  IL 6 blood level (ng/L) at the 1. Insertion of the retractor, 2. Begining of OLV 3. End of surgery, 4. Six hours after surgery

SECONDARY OUTCOMES:
IL8 | intraoperatively , 6 hours after surgery
  IL 8 (mg/L) blood level at the 1. Insertion of the retractor, 2. Begining of OLV 3. End of surgery, 4. Six hours after surgery
IL10 | intraoperatively , 6 hours after surgery
  IL 10 blood level (ng/L) at the 1. Insertion of the retractor, 2. Begining of OLV 3. End of surgery, 4. Six hours after surgery
CRP | 24 hours after surgery
  CRP blood level 24 hours after surgery
Oxygenation index | 6h after surgery
  pO2/FiO2
Lung infiltration | 6h after surgery
  X-ray of the lung- clear lungs, partly infiltrated lungs, totally infiltrated lungs

OTHER OUTCOMES:
Postoperative adverse events | 24h after surgery
  Prolonged antibiotics Pneumonia Reintubation SIRS ARDS Sepsis Death Acute Renal Failure Pooperative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Iztok Potocnik, MD, MSC, Principal Investigator — University Medical Centre Ljubljana; Vesna Novak Jankovic, MD, PROF, Study Chair — University Medical Centre Ljubljana
Locations (1):
- UMCLjubljana, CD of Anaesthesiology and Intensive Therapy, Ljubljana, Slovenia

REFERENCES:
- [Result] De Conno E, Steurer MP, Wittlinger M, Zalunardo MP, Weder W, Schneiter D, Schimmer RC, Klaghofer R, Neff TA, Schmid ER, Spahn DR, Z'graggen BR, Urner M, Beck-Schimmer B. Anesthetic-induced improvement of the inflammatory response to one-lung ventilation. Anesthesiology. 2009 Jun;110(6):1316-26. doi: 10.1097/ALN.0b013e3181a10731. PMID 19417610
- [Result] Schilling T, Kozian A, Senturk M, Huth C, Reinhold A, Hedenstierna G, Hachenberg T. Effects of volatile and intravenous anesthesia on the alveolar and systemic inflammatory response in thoracic surgical patients. Anesthesiology. 2011 Jul;115(1):65-74. doi: 10.1097/ALN.0b013e318214b9de. PMID 21399490
- [Result] Schilling T, Kozian A, Kretzschmar M, Huth C, Welte T, Buhling F, Hedenstierna G, Hachenberg T. Effects of propofol and desflurane anaesthesia on the alveolar inflammatory response to one-lung ventilation. Br J Anaesth. 2007 Sep;99(3):368-75. doi: 10.1093/bja/aem184. Epub 2007 Jul 9. PMID 17621602
- [Derived] Potocnik I, Novak Jankovic V, Sostaric M, Jerin A, Stupnik T, Skitek M, Markovic-Bozic J, Klokocovnik T. Antiinflammatory effect of sevoflurane in open lung surgery with one-lung ventilation. Croat Med J. 2014 Dec;55(6):628-37. doi: 10.3325/cmj.2014.55.628. PMID 25559834